CLINICAL TRIAL: NCT00248768
Title: Accelerated Transcranial Magnetic Stimulation for Depression
Brief Title: Accelerated Transcranial Magnetic Stimulation (TMS) for Depression
Acronym: ATMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3357-R; Emory IRB 601-2004 (Other: Emory IRB); NCT00449371 (obsolete NCT alias)
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Depression
Keywords: Depression; Parkinson Disease; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Other)
  Interventions: Device: Transcranial magnetic Stimulator

INTERVENTIONS:
Device: Transcranial magnetic Stimulator — a device which produces intense magnetic fields in the brain and activates cerebral neurons

SUMMARY:
The purpose of this study is to determinate if accelerated rTMS treatment over 1.5 days is effective for ameliorating depression in Parkinson's disease.

DETAILED DESCRIPTION:
Objective: The goal of this study is to investigate a new approach to administering repetitive transcranial magnetic stimulation (rTMS) in patients with refractory depression. (Please Note: The original requirement for comorbid Parkinson's disease has been dropped from this study).

Research Plan: This inpatient study will provide an initial test for the hypothesis that accelerated rTMS is an effective treatment for depression. Followup testing will help delineate the time course of response.

Methods: The rTMS treatment site over left dorsolateral prefrontal cortex will be 5.5cm anterior to the hand motor area. Treatments consisting of 1000 total pulses at 10 Hz and 100% motor threshold will be administered hourly for 1.5 days, totaling 15 sessions. A comprehensive test battery will be administered just before and after treatment, at 3 weeks, and at 6 weeks after treatment.

Clinical Relevance: We expect that accelerated rTMS treatments will lessen the degree of depression to the same extent as rTMS treatments of longer duration, but far more rapidly. A much shorter hospitalization would be more easily tolerated. In addition, reducing the duration of hospitalization substantially reduces burdens and costs to hospital, staff, and caregivers, while more rapidly enhancing function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Patients who meet DSM-IV criteria for Major Depressive Episode, severe, treatment resistant, with or without psychotic features.
* Consent to treatment with rTMS.

Exclusion Criteria:

* Patients with Delirium or Substance Dependence within the last 6 months. Patients will be screened initially with the Michigan Alcohol Screening Test (MAST) and Mini-Mental Status Examination and further evaluated if clinically indicated.
* Patients with other significant central neurological disorders including increased intracranial pressure, brain mass, epileptic seizures, stroke, transient ischemic attack within two years, cerebral aneurysm, dementia, multiple sclerosis or other major CNS dysfunction.
* Pregnant women.
* Patients with cardiac pacemakers, other intracardiac lines, cochlear implants, aneurism clips, or other intracranial implants with the exception of dental fillings.
* Patients with significant heart disease or with acute, unstable medical conditions that require stabilization (e.g., uncontrolled hypertension, bleeding) prior to treatment.
* Patients who require continued treatment with antipsychotics including clozapine and risperidone, benzodiazepines, lithium or anticonvulsants. Patients will be allowed to continue on a stable dose of antidepressants and use zolpidem, since the latter is not felt to affect seizure threshold.
* Patients who are unable to ambulate independently and complete the assessment protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale | 2-42 days

CONTACTS AND LOCATIONS:
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

REFERENCES:
- [Result] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360